CLINICAL TRIAL: NCT00023114
Title: p450 Mediated Lung Toxicity
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8408-CP-001
Record Dates: First submitted 2001-08-22; First posted 2001-08-24 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Pulmonary Disease
Keywords: lung function; smoking; metabolism
MeSH Terms: conditions — Lung Diseases; Smoking

SUMMARY:
The purpose of this project is to do cross species comparisons of the metabolism and toxicity of a number of toxicants which require metabolism for toxicity. All of the toxicants in question are encountered by humans in the workplace, through lifestyle choices (cigarette smoking) and as a result of environmental contamination. The high incidence of pulmonary diseases in the human population means that it will be difficult if not impossible to determine whether humans are at risk from exposure to these chemicals without solid mechanistic data. Recent rodent bioassays suggest that these compounds have oncogenic potential further supporting the need to test the potential for injury in primates. As part of this testing, we intend to establish in vitro methods for assessing critical steps in the metabolism of these agents and their interaction with cellular macromolecules. Once this is done, similar studies can be conducted in Rhesus or in human lung tissue that is available because it cannot be used for transplant purposes.

ELIGIBILITY:
All available organ donors in the Sacramento area

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2000-09; Study Completion 2001-09